CLINICAL TRIAL: NCT00006591
Title: The Safety and Efficacy of a Ritonavir-Enhanced Agenerase Regimen as Salvage Therapy in HIV-Infected Individuals
Brief Title: Ritonavir and Agenerase Treatment for Patients Who Have Failed Previous Anti-HIV Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gathe, Joseph, M.D. (Individual)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 313A; APV-430
Record Dates: First submitted 2000-12-01; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-12

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; VX 478; Salvage Therapy; Anti-HIV Agents; Drug Monitoring; Nelfinavir; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; amprenavir

INTERVENTIONS:
Drug: Ritonavir
Drug: Amprenavir

SUMMARY:
The purpose of this study is to determine if treatment with an anti-HIV drug containing ritonavir and Agenerase is safe and can lower the level of HIV in the blood in patients who have failed an anti-HIV drug treatment containing nelfinavir.

DETAILED DESCRIPTION:
HIV-infected patients will be treated with a ritonavir-enhanced Agenerase regimen.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 18 years of age or older.
* Are HIV-positive.
* Have a viral load (level of HIV in the body) of more than 1,000 copies/ml.
* Have had more than 12 weeks of prior anti-HIV drug treatment.
* Have failed a previous anti-HIV treatment containing nelfinavir as the only protease inhibitor.
* Are responsive to Agenerase.
* Are able to follow study requirements.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are intolerant to ritonavir (an anti-HIV drug).
* Have or have had problems with absorption.
* Have liver disease or damage.
* Have pancreatic disease or damage.
* Have taken any protease inhibitor other than nelfinavir.
* Are receiving investigational drugs or devices from another study.
* Are pregnant or breast-feeding.
* Currently use triazolam, astemizole, ergot medications, cisapride, midazolam, bepridil, rifampin, terfenadine, or pimozide.
* Have a bleeding disorder.
* Have previously been treated with Agenerase.
* Are receiving nonnucleosides.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Gathe, Joseph, M.D., Houston, Texas, United States